CLINICAL TRIAL: NCT01026155
Title: Respiratory Muscle Endurance Training in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Edith Seltzer (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Respob
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Obesity
Keywords: Obese patients (BMI > 30 kg / m²)
MeSH Terms: conditions — Obesity | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory muscle traininig (Experimental): Low caloric diet and physical activities + Respiratory muscle endurance training by means of isocapnic voluntary hyperpnoea
  Interventions: Other: Respiratory muscle training
- Control (Active Comparator): Low caloric diet and physical activities
  Interventions: Other: Respiratory muscle training

INTERVENTIONS:
Other: Respiratory muscle training — Respiratory muscle endurance training by means of isocapnic voluntary hyperpnoea

SUMMARY:
Obese patients are known to have increased work of breathing inducing dyspnea, exercise intolerance and impaired quality of life. Respiratory muscle training is known to increase respiratory muscle capacity, reduce dyspnoea and improve exercise performance in healthy subjects and respiratory patients. The investigators hypothesized that Respiratory muscle training would reduce dyspnoea, increase exercise tolerance and quality of life in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI > 30 kg/m2), without respiratory pathology (VEMS > 80% predicted, VEMS/CV > 80%)
* men or women
* age between 18 and 60 years old

Exclusion Criteria:

* Respiratory, cardiovascular, musculoskeletal diseases
* Alcoholism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)

PRIMARY OUTCOMES:
Dyspnea at rest and during exercise

SECONDARY OUTCOMES:
Exercise performance (6-min walking distance) Quality of life (SF36 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wuyam, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Centre Bois de l'Ours, Briançon, France